CLINICAL TRIAL: NCT05828537
Title: the Use of PEDI_EAT 10 Score Versus Nurse Performed Screening in the Assessment of Post Extubation Dysphagia
Brief Title: The Use of PEDI_ EAT 10 Score Versus Nurse Performed Screening in the Assessment of Post Extubation Dysphagia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gaber Hassaan Mohamed, resident, Assiut University
Other Study IDs: pedi postextubation dysphagia
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pediatric Post Extubation Dysphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endotracheal tube — pediatric extubation

SUMMARY:
Invasive mechanical ventilation is one of the most common interventions in critically ill patients, and is invariably characteristic, if not defining, of ICU therapeutic regimen Much attention has been paid to complications occurring during and because of mechanical ventilation, such as nosocomial infections, delirium, and critical illness neuropathy and myopathy. However, an often underappreciated and minimally explored complication of mechanical ventilation is post-extubation dysphagia .

DETAILED DESCRIPTION:
Invasive mechanical ventilation is one of the most common interventions in critically ill patients, and is invariably characteristic, if not defining, of ICU therapeutic regimen Much attention has been paid to complications occurring during and because of mechanical ventilation, such as nosocomial infections, delirium, and critical illness neuropathy and myopathy. However, an often underappreciated and minimally explored complication of mechanical ventilation is post-extubation dysphagia .

Post-extubation dysphagia (PED) is defined as the difficulty or inability to effectively and safely transfer food and liquid from the mouth to the stomach after extubation.

As reported by Malandraki et al PED is more common in pediatric patients with an overall incidence of 29% and exceeds the 23% incidence reported in adults, Another Australian context showed that 41% of critically-ill pediatric patients requiring endotracheal intubation eventually evolved PED with one-third of those patients experiencing silent aspiration.

Using a prior pioneering prospective study of mechanically ventilated patients, Zuercher et al evaluated 933 extubated patients, of which 116 were screened for the presence of post-extubation dysphagia. They analyzed pre-intubation characteristics to derive factors possibly associated with development of PED, and found that pre-existing neurological disease, emergency admission, increased duration of mechanical ventilation, increased duration of renal replacement therapy, and higher severity of illness were associated with development of post- extubation dysphagia. Interestingly, increased BMI was associated with lower incidence of dysphagia.

Because of the significant negative impact of post-extubation dysphagia on outcomes of pediatric patients, early identification and intervention are crucial. The scientific description of the phenomenon of post-extubation dysphagia in pediatric populations as a distinct pathological entity from the phenomenon in adult populations is considered a corner stone in the systematic exploration of the phenomenon . Such systematic exploration has, to date, been limited...

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients admitted to PICU and needed mechanical ventilation

Exclusion Criteria:

* patient admitted to PICU but not neeed MV

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pediatric patients admitted to PICU and needed MV
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the efficiency of PED EAT 10 tool versus nurse performed screening to reliably evaluate PED among all ICU patients needed mechanical ventilation by detecting outcome: -oral feeding at ICU discharge | 1 year
  Assessing the efficiency of PED EAT 10 tool versus nurse performed screening to reliably evaluate PED among all ICU patients needed mechanical ventilation by detecting outcome:
  -oral feeding at ICU discharge

SECONDARY OUTCOMES:
Assessing the efficiency of PED EAT 10 tool versus nurse performed screening to reliably evaluate PED among all ICU patients needed mechanical ventilation by detecting outcome: ICU readmission. | 1 year
  Assessing the efficiency of PED EAT 10 tool versus nurse performed screening to reliably evaluate PED among all ICU patients needed mechanical ventilation by detecting outcome:
  ICU readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Azhar A Mohamed, lecturer, Study Director — Assiut University